CLINICAL TRIAL: NCT00054977
Title: A Phase I Open-Label Study to Evaluate the Safety and Tolerability of Escalating Doses of GM-CT-01 in the Presence and Absence of 5-Fluorouracil (5-FU) in Subjects With Advanced Solid Tumors
Brief Title: Safety of GM-CT-01 With and Without 5-Fluorouracil in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galectin Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAVFU-001
Record Dates: First submitted 2003-02-14; First posted 2003-02-17 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Colorectal Cancer; Lung Cancer; Breast Cancer; Head and Neck Cancer; Prostate Cancer
Keywords: cancer; tumor
MeSH Terms: conditions — Colorectal Neoplasms; Lung Neoplasms; Breast Neoplasms; Head and Neck Neoplasms; Prostatic Neoplasms; Neoplasms | interventions — galactomannan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GM-CT-01 — IV infusion over 30 minutes of 6 Dosages escalated from 30 to 280 mg/m2, given for 4 consecutive days in a 28 days cycle.
  Other Names: DAVANAT
Drug: 5-fluorouracil — IV infusion over 30 minutes at Dosage of 500 mg/m2, given in-combination with GM-CT-01, for 4 consecutive days in a 28 days cycle.
  Other Names: 5-FU

SUMMARY:
This is a Phase I, multi-center study of GM-CT-01, which has been shown to increase the anti-tumor activity of 5-fluorouracil in mice. The primary reason for doing the study is to determine the safety of GM-CT-01 given alone and in combination with therapeutical dosage of 5-Fluorouracil, in patients who have advanced cancer that can be measured by CT scan.

DETAILED DESCRIPTION:
5-Fluorouracil is a chemotherapy drug commonly used in cancer patients. Patients with different type of solid tumors who have failed standard, approved treatments can be enrolled in the study. Escalated doses of GM-CT-01 will be given alone in Cycle 1, and in combination with 5-fluorouracil in cycle 2. Patients will be on study for approximately 60 days for determination of safety. However, with patient consent treatment can continue until disease progression is determined by CT scan. The study secondary reason is to determine whether treatment has stabilize the tumors or change it in size (get bigger, smaller or stay the same)after Cycle 2 and any additional cycles of treatment.

ELIGIBILITY:
Inclusion Criteria:

* The subject is able to give informed consent to participate in this trial (including all procedures and follow-up visits).
* The subject is male or female at least 18 years of age.
* The subject has a documented histologic or cytologic recurrent or metastatic solid tumor that is not amenable to curative surgery, radiotherapy, or conventional chemotherapy of proven value.
* Subjects must have completed previous therapy (chemotherapeutic agents or other therapies including radiation) at least 4 weeks prior to study entry.
* Following major surgery (e.g. laparotomy), > 4 weeks must have elapsed and subjects must have recovered from effects.
* Following minor surgery (does not include insertion of vascular access device), > 2 weeks must have elapsed.
* ECOG performance status of 0-2.
* The subject has a life expectancy of at least 12 weeks.
* Female subjects must be post-menopausal, surgically sterile, or using effective contraception.

Laboratory values prior to administration of study drug:

* If female and not post-menopausal, the subject has a negative pregnancy test.
* Liver function studies: AST and ALT < 2.5 times the upper limit of normal (ULN); total bilirubin < 1.5
* Hematopoietic parameters: WBC > 3000 per mm3; Granulocyte count > 1,500 per mm3; Platelet count > 100,000 per mm3
* Renal: Creatinine < or = ULN
* Pulmonary: Dlco > or = 60% of predicted

Exclusion Criteria:

* If female, the subject is pregnant or breast feeding.
* Central nervous system (CNS) metastases or primary CNS tumors.
* The subject has a known hypersensitivity to GM-CT-01 or any of its components.
* The subject has congestive heart failure or any other medical condition that could be adversely affected by intravenous infusion of up to approximately 200 mL of fluid over 60 minutes.
* The subject is currently abusing alcohol and/or illicit drugs.
* The subject has other significant medical, psychiatric, or social conditions which, in the investigators' opinion, may compromise the subject's safety in participating in this study.
* In the investigators' judgment, the subject would be unreliable in adhering to the study visit schedule or other study requirements.
* The subject is currently enrolled in a clinical trial or has participated in a clinical trial within the 30 days prior to entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2003-02; Primary Completion 2005-04 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Safety | 60 days - two cycles of treatment

SECONDARY OUTCOMES:
Tumor progression | CT imaging at 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn C Pike, M.D., Ph.D., Study Director — Consultant to Pro-Pharmaceuticals, Inc.
Locations (4):
- United States (4):
  - Florida Oncology Associates, Jacksonville, Florida
  - Ochsner Cancer Institute, New Orleans, Louisiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire